CLINICAL TRIAL: NCT07079228
Title: A Phase 3, Multi-Center, Double-blind, Randomized Study of QLS31905 Plus Chemotherapy Versus Placebo Plus Chemotherapy as First-Line Treatment in Participants With Claudin (CLDN)18.2-Positive Advanced Pancreatic Cancer
Brief Title: A Study to Compare QLS31905 and Chemotherapy With Placebo and Chemotherapy in Participants With Pancreatic Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QLS31905-301
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLS31905 + nab-paclitaxel + gemcitabine (AG) (Experimental)
  Interventions: Drug: QLS31905; Drug: Nab-paclitaxel.; Drug: Gemcitabine
- Placebo + nab-paclitaxel + gemcitabine (AG) (Active Comparator)
  Interventions: Drug: Placebo for QLS31905; Drug: Nab-paclitaxel.; Drug: Gemcitabine

INTERVENTIONS:
Drug: QLS31905 — QLS31905 will be administered as an IV infusion.
  Arms: QLS31905 + nab-paclitaxel + gemcitabine (AG)
Drug: Nab-paclitaxel. — Nab-paclitaxel will be administered as an IV infusion.
  Arms: QLS31905 + nab-paclitaxel + gemcitabine (AG)
Drug: Gemcitabine — Gemcitabine will be administered as an IV infusion.
  Arms: QLS31905 + nab-paclitaxel + gemcitabine (AG)
Drug: Placebo for QLS31905 — Placebo will be administered as an IV infusion.
  Arms: Placebo + nab-paclitaxel + gemcitabine (AG)
Drug: Nab-paclitaxel. — Nab-paclitaxel will be administered as an IV infusion
  Arms: Placebo + nab-paclitaxel + gemcitabine (AG)
Drug: Gemcitabine — Gemcitabine will be administered as an IV infusion.
  Arms: Placebo + nab-paclitaxel + gemcitabine (AG)

SUMMARY:
The goal of this study is to evaluate the efficacy of QLS31905 in combination with chemotherapy (nab-paclitaxel plus gemcitabine [AG]) versus placebo in combination with chemotherapy (AG) in the treatment of CLDN18.2-positive advanced pancreatic cancer in adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in the study and sign the informed consent form;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
* Expected survival time ≥ 3 months;
* Histologically or cytologically confirmed diagnosis of pancreatic cancer;
* No prior systemic anti-tumor treatment for unresectable locally advanced or metastatic disease;
* At least one measurable lesion per RECIST v1.1;
* Patients with adequate cardiac, liver, renal function, etc.

Exclusion Criteria:

* History of malignancies other than the target cancer within 5 years prior to the first dose of the investigational product ;
* Underwent major organ surgery (excluding needle biopsy) or had significant trauma within 28 days prior to enrollment, or requires elective surgery during the study;
* Known central nervous system metastases;
* Patients with hepatitis B; patients with hepatitis C; patients who test positive for syphilis, or patients with a known history of HIV or positive HIV screening test;
* Patients with added risks associated with the study or may interfere with the interpretation of study results as determined by the investigator, or deemed unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Overall Suryival(OS) | Up to 48 months
  OS is defined as the time from randomization to deathdue to any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 48 months
  PFS is defined as the duration from randomization to the first imaging confirmation of progressive disease per RECIST 1.1 by investigator evaluation or death due to any cause (whichever occurs first).
Objective Response Rate (ORR) | Up to 48 months
  ORR is defined as the proportion of participants who have a best overall response of Complete Response (CR) or Partial Response (PR) as assessed by investigator evaluation per RECIST 1.1.
  Time Frame: Up to 48 months
Duration Of Response (DOR) | Up to 48 months
  DOR is defined as the time from the date of the first response (CR/PR) until the date of progressive disease as assessed by investigator evaluation per RECIST 1.1 or death due to any cause (whichever occurs first).
Safety assessed by Adverse Events (AEs) | Up to 48 months
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom,or disease (new or exacerbated) temporally associated with the use of a medicinal product.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China